CLINICAL TRIAL: NCT05770518
Title: Biofeedback vs Laryngeal Control Therapy in Management of Paradoxical Vocal Fold Motion (BLiMP)
Brief Title: Biofeedback vs Laryngeal Control Therapy in Management of Paradoxical Vocal Fold Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202210154
Record Dates: First submitted 2023-03-02; First posted 2023-03-15 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Paradoxical Vocal Fold Motion; Vocal Cord Dysfunction
Keywords: laryngeal control therapy; biofeedback; dyspnea; stridor; dysphonia; cough; laryngoscopy
MeSH Terms: conditions — Vocal Cord Dysfunction; Dyspnea; Respiratory Sounds; Dysphonia; Cough | interventions — Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: Pilot randomized controlled trial with active treatment control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback (Experimental): In office video biofeedback performed at the time of the diagnosis.
  Interventions: Behavioral: Biofeedback
- Laryngeal control therapy (Active Comparator): A specific type of behavioral therapy performed by speech and language pathologists
  Interventions: Behavioral: Laryngeal control therapy (LCT)

INTERVENTIONS:
Behavioral: Biofeedback — Biofeedback is a strategy used in the treatment of PVFM, which involves allowing patients to directly visualize their breathing patterns during laryngoscopy.
  Other Names: Video biofeedback
  Arms: Biofeedback
Behavioral: Laryngeal control therapy (LCT) — This treatment typically involves 2 guided therapy sessions that include patient education, relaxation techniques, and training in specific breathing techniques.
  Other Names: respiratory retraining
  Arms: Laryngeal control therapy

SUMMARY:
Paradoxical Vocal Fold Motion (PVFM) is a condition where vocal cords adduct (move toward another) instead of abduct (move away from one another) during inspiration, thus causing shortness of breath. The goal of this pilot randomized controlled trial is to compare the efficacy of biofeedback as compared to laryngeal control therapy (LCT) in the treatment of PVFM. Participants will take surveys about their symptoms and their expectations of treatment prior to initiating treatment and after completion of their assigned treatment. Researchers will compare the biofeedback group to the LCT group to see if participants have differences in changes of their symptoms.

DETAILED DESCRIPTION:
Paradoxical vocal fold motion (PVFM) is characterized by episodic shortness of breath that can range in severity and acuity. Symptoms may greatly impact daily life. Some patients experience severe respiratory distress, which can lead to emergency department visits and occasionally intubation. The standard treatment is typically behavioral therapy performed by speech and language pathologists. However, new evidence suggests that video biofeedback may be an effective alternative treatment. Video biofeedback allows patients to directly visualize their breathing while performing specific breathing exercises. This is a desirable treatment because it can be performed at the time of diagnosis and requires minimal additional time or resources. The investigators' goal is to conduct a pilot randomized controlled trial (RCT) to compare the relative effectiveness of video biofeedback and behavioral therapy in the treatment of PVFM. The primary endpoint will be the change in Dyspnea Index score before treatment and one month after treatment. Patients will complete surveys to collate data about patient expectations of behavioral therapy, their reasons for pursuing additional treatment if applicable, and the perceived benefits of the specific intervention. The investigators hypothesize that no clinically meaningful difference will be detected between behavioral therapy and video biofeedback for the treatment of PVFM. This pilot RCT will provide critical data for designing a fully powered trial comparing these two interventions, and will advance the investigators' goal of providing clinicians with important evidence for guiding treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or older
* Referral to the Washington University School of Medicine Voice and Airway Center for concerns for PVFM
* Pre-treatment Dyspnea Index score of 11 or higher (representing the threshold for having an abnormal score)
* Answer yes to the following questions: "Do you sometimes have difficulty breathing?" and "When you have difficulty breathing, is it worse when inhaling (breathing in)?"

Exclusion Criteria:

* Inability to speak or understand English
* Previous treatment of PVFM
* History of laryngeal surgery
* Evidence of alternative laryngeal pathology (e.g. subglottic stenosis, benign or malignant obstructive mass) on flexible laryngoscopy as performed as part of routine clinical care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Dyspnea Index (DI) | pre and 1 month post treatment
  This is a 10-item questionnaire with scores that range from 0-40, with 40 representing the greatest possible severity of symptoms.
  The DI is a clinical assessment tool that was designed and validated specifically for patients with upper airway obstruction, including patients with PVFM.
  The primary outcome measure will be the difference between the two groups in the change in Dyspnea Index (DI).

SECONDARY OUTCOMES:
Dyspnea Index (DI) | pre and 3 months post treatment
  This is a 10-item questionnaire with scores that range from 0-40, with 40 representing the greatest possible severity of symptoms.
  The DI is a clinical assessment tool that was designed and validated specifically for patients with upper airway obstruction, including patients with PVFM.
  The primary outcome measure will be the difference between the two groups in the change in Dyspnea Index (DI).
Responder rates | 1 month and 3 months post treatment
  Responder rate is the proportion of subjects at 1 month post-treatment whose Dyspnea Index scores have decreased by at least the minimal clinically important difference.
The Clinical Global Impressions - Improvement (CGI-I) | 1 month and 3 months post treatment
  This is a widely used research rating tool which will be used to assess the response to treatment using a 7-point Likert scale. A score of 1 represents maximal improvement of symptoms, and a score of 7 represents maximal worsening of symptoms. Language has been adapted to represent participants' changes in breathing quality.
Qualitative Survey | 3 months post treatment
  The investigators will ask participants questions about their expectations of treatment, reasons for pursuing additional treatment if applicable, and perceived utility of their treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Huston, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George S, Suresh S. Vocal Cord Dysfunction: Analysis of 27 Cases and Updated Review of Pathophysiology & Management. Int Arch Otorhinolaryngol. 2019 Apr;23(2):125-130. doi: 10.1055/s-0038-1661358. Epub 2018 Oct 24. PMID 30956693
- [Background] Kramer S, deSilva B, Forrest LA, Matrka L. Does treatment of paradoxical vocal fold movement disorder decrease asthma medication use? Laryngoscope. 2017 Jul;127(7):1531-1537. doi: 10.1002/lary.26416. Epub 2016 Nov 15. PMID 27861929
- [Background] Guglani L, Atkinson S, Hosanagar A, Guglani L. A systematic review of psychological interventions for adult and pediatric patients with vocal cord dysfunction. Front Pediatr. 2014 Aug 8;2:82. doi: 10.3389/fped.2014.00082. eCollection 2014. PMID 25152871
- [Background] Mahoney J, Hew M, Vertigan A, Oates J. Treatment effectiveness for Vocal Cord Dysfunction in adults and adolescents: A systematic review. Clin Exp Allergy. 2022 Mar;52(3):387-404. doi: 10.1111/cea.14036. Epub 2021 Nov 4. PMID 34699093
- [Background] Shaffer M, Litts JK, Nauman E, Haines J. Speech-Language Pathology as a Primary Treatment for Exercise-Induced Laryngeal Obstruction. Immunol Allergy Clin North Am. 2018 May;38(2):293-302. doi: 10.1016/j.iac.2018.01.003. Epub 2018 Mar 2. PMID 29631737
- [Background] Patel RR, Venediktov R, Schooling T, Wang B. Evidence-Based Systematic Review: Effects of Speech-Language Pathology Treatment for Individuals With Paradoxical Vocal Fold Motion. Am J Speech Lang Pathol. 2015 Aug;24(3):566-84. doi: 10.1044/2015_AJSLP-14-0120. PMID 25836980
- [Background] Gartner-Schmidt JL, Shembel AC, Zullo TG, Rosen CA. Development and validation of the Dyspnea Index (DI): a severity index for upper airway-related dyspnea. J Voice. 2014 Nov;28(6):775-82. doi: 10.1016/j.jvoice.2013.12.017. Epub 2014 Oct 12. PMID 25311596
- [Background] LeBlanc RA, Aalto D, Jeffery CC. Visual biofeedback for paradoxical vocal fold motion (PVFM). J Otolaryngol Head Neck Surg. 2021 Feb 18;50(1):13. doi: 10.1186/s40463-021-00495-0. PMID 33602342
- [Background] De Guzman V, Ballif CL, Maurer R, Hartnick CJ, Raol N. Validation of the dyspnea index in adolescents with exercise-induced paradoxical vocal fold motion. JAMA Otolaryngol Head Neck Surg. 2014 Sep;140(9):823-8. doi: 10.1001/jamaoto.2014.1405. PMID 25104182
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Derived] Strober WA, Rohlfing ML, Cutchin GM, Kallogjeri D, Piccirillo JF, Huston MN. Biofeedback vs Respiratory Retraining for Inducible Laryngeal Obstruction: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2025 Dec 11:e254542. doi: 10.1001/jamaoto.2025.4542. Online ahead of print. PMID 41379457